CLINICAL TRIAL: NCT02465723
Title: Detection of Acid Sphingomyelinase/Ceramide Pathway Activation in Radiotherapy Patients Using Intravoxel Incoherent Motion (IVIM) Diffusion-weighted Magnetic Resonance Imaging and Serum Biomarkers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-104
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Metastatic Disease to Bone; Metastatic Disease to Soft Tissue
Keywords: Intravoxel Incoherent Motion (IVIM); Diffusion-weighted Magnetic Resonance; Acid Sphingomyelinase/Ceramide Pathway Activation; 15-104
MeSH Terms: interventions — Blood Specimen Collection

ARMS (1):
- MRI with IVIM DW-MRI (Experimental): Upon enrollment in the study, each patient will undergo a standard pre-treatment evaluation in the Radiation Oncology Clinic. Imaging will include MRI with IVIM DW-MRI (as a research exam). MR imaging will begin within 30 minutes (+/- 15 mins) of the completion of single-dose radiation or the first dose for patients treated with a multifractioned regime. Patients will have corresponding serum samples collected at approximately 1 hour before and 18-24 hours after the first radiation treatment. If radiation therapy occurs on a Friday, the collection of the serum 18-24 hours post-treatment may still be feasible. Patients will be treated with radiation therapy according to our standard clinical guidelines using one of several Varian megavoltage linear accelerators with on-board kilovoltage image-guidance capabilities, using established immobilization devices that are specific to the anatomical site treated at MD's discretion.
  Interventions: Device: MRI with IVIM DW-MRI; Other: Blood draw

INTERVENTIONS:
Device: MRI with IVIM DW-MRI
Other: Blood draw — For each patient enrolled, 8-10 mL of whole blood will be collected into glass, anti-coagulant-free tubes and allowed to clot 20-30 minutes.

SUMMARY:
The purpose of this study is to find out if special blood tests and imaging scans can help evaluate the effects of the radiation the patient receives as part of standard treatment. The patient will undergo either stereotactic or conventional radiation treatment as determined by the treating doctor. Previous evidence suggests that blood flow to tumors is affected by the amount (dose) of radiation that it receives. This effect may be seen as soon as 1-2 hours after the radiation is given. This study will evaluate if these changes can be seen and measured by performing a special type of scan called Intravoxel Incoherent Motion (IVIM) diffusion-weighted Magnetic Resonance Imaging (MRI) and a blood test. IVIM MRI is a research exam which is similar to a standard MRI exam, with only a slight difference in the technical parameters used to acquire the images.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cancer
* Patients deemed clinically appropriate for radiation treatment as part of the standard care provided by their treating physician, and will receive either 24 Gy (one fraction) or 3 Gy x 10 fractions.
* Life expectancy > 6 months
* KPS>60%
* Age ≥ 18 years old.

Exclusion Criteria:

* Pregnant patients
* Patients who are unwilling or unable to undergo MRI including patients with contraindications to MRI such as the presence of cardiac pacemakers or non-compatible intracranial vascular clips, claustrophobia, inability to lie flat for the duration of the study etc
* Prior radiotherapy to the site of intended treatment
* Patients with tumor involving brain or spinal cord
* Platelet count <75,000/μl, HgB level <9 g/dl, WBC <3500/μl
* Presence of metastases in the upper thoracic spine (in order to avoid DW- MRI parameter measurement variability due to cardiac motion)
* Lesions <1.5 cm (to assure robust measurements)
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
ASMase activity measurement | up to 18-24 hours after the first radiation treatment
  For each serum ASMase activity measurement, we will use 3 technical assay replicates. Each of three replicates will be averaged. Then the post-treatment activity will be normalized (fraction) against its paired pre-treatment activity.

SECONDARY OUTCOMES:
C16 serum ceramide levels | 1 year
  Total C16 serum ceramide level, expressed as ng of ceramide per mL, will be measured for the pre-RT serum and post-RT serum. For each patient, the post-RT C16 ceramide level will be expressed as a fraction of the pre-RT levels.
C18 serum ceramide levels | 1 year
  Total C18 serum ceramide level, expressed as ng of ceramide per mL, will be measured for the pre-RT serum and post-RT serum. For each patient, the post-RT C18 ceramide level will be expressed as a fraction of the pre-RT levels.

CONTACTS AND LOCATIONS:
Overall Officials: Hebert A. Vargas, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/